CLINICAL TRIAL: NCT00340314
Title: A Controlled Randomized Trial of Circumferential Pulmonary Vein Ablation Versus Antiarrhythmic Drug Therapy in Treating Paroxysmal Atrial Fibrillation. The Ablation for Paroxysmal Atrial Fibrillation (APAF2) Trial
Brief Title: A Trial of Circumferential Pulmonary Vein Ablation (CPVA) Versus Antiarrhythmic Drug Therapy in for Paroxysmal Atrial Fibrillation (AF)
Acronym: APAF2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APAF/02
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2006-05

CONDITIONS: Atrial Fibrillation
Keywords: symptomatic; paroxysmal; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

INTERVENTIONS:
Procedure: Circumferential Pulmonary Vein Ablation
Drug: Antiarrhythmic Drug Therapy

SUMMARY:
Background: Circumferential pulmonary vein ablation (CPVA) has been safely and effectively performed for treating paroxysmal atrial fibrillation (PAF); however, its safety and efficacy, as compared with those of antiarrhythmic drug therapy (ADT), have never been formally assessed in a randomized controlled trial.

The Purpose of this study was to evaluate CPVA versus ADT in patients with PAF in a randomized controlled trial.

DETAILED DESCRIPTION:
Antiarrhythmic drug therapy (ADT) is currently considered as first-line therapy in patients with paroxysmal atrial fibrillation (AF).1 However antiarrhythmic drugs are frequently ineffective and can have serious potential adverse effects, thus often offsetting any advantage offered by the maintenance of sinus rhythm (SR).2,3 Data from our and other laboratories suggest that pulmonary vein ablation techniques may be a curative alternative for AF, obviating the need for ADT and/or anticoagulation in many patients.4-8 However, only preliminary and frequently non-randomized data exists for an evidence-based evaluation of catheter ablation as compared to conventional antiarrhythmic drug therapyADT.4,8 Thus, we conducted a controlled randomized trial (the Ablation for Paroxysmal Atrial Fibrillation [APAF] trial) to determine the long-term efficacy of circumferential pulmonary vein ablation (CPVA) in patients with paroxysmal AF as compared with ADT with flecainide, sotalol or amiodarone.

Methods: One hundred ninety-eight patients (age, 56±10 years) with PAF (duration, 6±5 years, mean AF episodes 3.4/month), were randomized to CPVA or to ADT with flecainide, sotalol or amiodarone. Ablation was randomly performed with the use of a standard or an irrigated tip catheter and with CARTO or NavX non fluoroscopic 3D systems guidance. Cardiac rhythm was assessed with daily transtelephonic transmissions over a 12 and 48 months follow-up. Crossovers to CPVA were allowed after 3 months of ADT.

Results: By Kaplan-Meier analysis, 86% of patients in the CPVA group and 22% in the ADT group were free from recurrent atrial tachyarrhythmias ([AT] P<0.001); a repeat ablation was performed in 9% of patients in the CPVA group for recurrent AF (6%) or atrial tachycardia (3%). At 1 year, 93% and 35% of the CPVA and ADT groups were AT-free while at 4 years only 72.7% patients assigned to RFA and 12.1% assigned to AADs reached the endpoint(p<0.001).Lower left ejection fraction, arterial hypertension and age independently predicted AF recurrences in the ADT group. CPVA was associated with a significant decrease in left atrial diameter (15±10%, P<0.01) and with fewer number of cardiovascular hospitalizations (p<0.01). Ablation with an irrigated tip catheter was more effective (P=0.03) with either the CARTO or NavX system (P=0.08). One transient ischemic attack and one pericardial effusion occurred in the CPVA group; side effects of ADT were reported in 23 patients.During the 4-year follow-up, 87 initially AADs patients required cross over to RFA with a steeper rate at 1 year (42 patients) and 19 of them progressed to persistent AF before switching. Considering repeat ablation and crossover, the overall success rate was 90% in RFA group and 80% in AAD group (p=0.0023, by log-rank test). New left AT developed in 9 patients requiring mapping and ablation in 7 patients. Quality of life was higher in the RFA group than in AAD group for all subscale scores (p<0.001) Conclusions: Compared to ADT, CPVA can safely and effectively cure PAF in many patients at one-year follow-up and this benefit is extended to 4 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years
2. History of symptomatic paroxysmal AF lasting more than 6 months. Paroxysms of AF are intended as recurrent self-terminating episodes lasting less than 7 days and occurring more than 2 times every month.

Exclusion Criteria:

1. Pregnancy
2. NYHA functional class III or IV
3. Left atrial size > 65 mm
4. Left ventricular (LV) ejection fraction < 35%
5. Contraindication to anticoagulation with warfarin
6. History of myocardial infarction within six months of the procedure
7. Prior catheter or surgical ablation attempt for AF
8. Inability or unwillingness to provide written informed consent
9. Life expectancy less than 1 year
10. Significant comorbid conditions such as: cancer (not cured), end stage renal disease (creatinine clearance < 20 mL/h), severe chronic obstructive lung disease, cirrhosis, etc)
11. Anticipated cardiac surgery for congenital, valvular, aortic or coronary heart disease.
12. Presence of left atrial thrombus.
13. Prior antiarrhythmic drug therapy with amiodarone, sotalol and flecainide at optimal doses (target 200 mg, 240 mg, 200 mg daily respectively
14. AF burden < 2 episodes/month
15. WPW
16. Expected survival < 1 year
17. Contraindications for antiarrhythmics therapy including flecainide, sotalol or amiodarone not listed above:

    * LV hypertrophy (LV mass index > 125g/m2)
    * thyroid dysfunction (hyperthyroidism or uncontrolled hypothyroidism or thyroid cancer)
    * liver dysfunction (ALT or AST >2x the reference values)
    * Interstitial lung disease with DLCO<70% of predicted or severe asthma.
    * QT interval exceeding 400 msec
    * Symptomatic sinus node or atrioventricular node dysfunction unless a pacemaker had been implanted
    * Evidence of stress-induced myocardial ischemia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198
Dates: Start 2005-01; Study Completion 2006-05

PRIMARY OUTCOMES:
The primary end point was freedom from recurrent atrial tachyarrhythmias ([AT], both AF and regular atrial tachycardia) during a 12 and 48 months follow-up . The first analysis was scheduled to be performed after the last enrolled patient complete.

SECONDARY OUTCOMES:
Presence of SR during 1-month intervals
Percent of patients totally free of AF
Number of cardioversions
LV function
Incidence of cardiovascular hospitalization
Overall morbidity
Left atrial size and function
Thromboembolic and bleeding complications
Efficacy and safety of two 3D mapping systems
Efficacy and safety of two ablation catheters
Procedure duration, length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Pappone, MD, PhD, Principal Investigator — San Raffaele University Hospital, Villa Maria Cecilia Hospital, Cotignola (Ravenna), Italy; Vincenzo Santinelli, MD, Study Chair — San Raffaele University Hospital, Villa Maria Cecilia Hospital, Cotignola (Ravenna), Italy
Locations (1):
- San Raffaele University Hospital, Milan, Italy

REFERENCES:
- [Derived] Pappone C, Vicedomini G, Augello G, Manguso F, Saviano M, Baldi M, Petretta A, Giannelli L, Calovic Z, Guluta V, Tavazzi L, Santinelli V. Radiofrequency catheter ablation and antiarrhythmic drug therapy: a prospective, randomized, 4-year follow-up trial: the APAF study. Circ Arrhythm Electrophysiol. 2011 Dec;4(6):808-14. doi: 10.1161/CIRCEP.111.966408. Epub 2011 Sep 23. PMID 21946315
- [Derived] Pappone C, Augello G, Sala S, Gugliotta F, Vicedomini G, Gulletta S, Paglino G, Mazzone P, Sora N, Greiss I, Santagostino A, LiVolsi L, Pappone N, Radinovic A, Manguso F, Santinelli V. A randomized trial of circumferential pulmonary vein ablation versus antiarrhythmic drug therapy in paroxysmal atrial fibrillation: the APAF Study. J Am Coll Cardiol. 2006 Dec 5;48(11):2340-7. doi: 10.1016/j.jacc.2006.08.037. Epub 2006 Oct 16. PMID 17161267
- See also: Our Departement Web site — http://www.af-ablation.org